CLINICAL TRIAL: NCT03213639
Title: Use of Esomeprazole in Treatment of Early Onset Preeclampsia:a Double Blind Randomized, Placebo-controlled Trial
Brief Title: Esomeprazole in Treatment of Early Onset Preeclampsia (ESOPE Trial)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ESOPE
Record Dates: First submitted 2017-07-08; First posted 2017-07-11 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Esomeprazole; Tablets; Noble Gases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Patients will take esomeprazole single dose of 40 mg orally once a day
  Interventions: Drug: Esomeprazole 40 mg Oral Tablet
- control group (Placebo Comparator): Patients will take an inert tablet similar in appearance, color and consistency
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Esomeprazole 40 mg Oral Tablet — once daily oral tablets
  Other Names: Nexium
  Arms: study group
Drug: Placebo Oral Tablet — once daily oral tablets
  Other Names: inert
  Arms: control group

SUMMARY:
Pre-eclampsia is one of the most serious complications of pregnancy affecting 3-8 % of pregnancies worldwide. It is a multi-system disorder involving maternal vessels (causing hypertension and endothelial dysfunction), the kidneys, the liver, the lungs, the hematological system, the cardiovascular system and the feto-placental unit. In its most severe form, it affects the brain, causing seizures (eclampsia), cerebro-vascular events and even death.

DETAILED DESCRIPTION:
The key aspects in the pathophysiology of pre-eclampsia are placental oxidative stress (and hypoxia), placental release of the anti-angiogenic factors Soluble Fms Like Tyrosine Kinase -1 and soluble endoglin and maternal endothelial dysfunction. A drug that can counter these pathological steps could be a strategy to treat pre-eclampsia.

If an affordable and safe treatment was available it could temporize the disease progression of pre-eclampsia thereby delaying delivery to gain gestation. This could save the lives of many infants and decrease the hospital burden caused by iatrogenic prematurity.

Currently, there are trials investigating the possible use of pravastatin to treat pre-eclampsia, and to prevent it There are no other significant trials of orally available small molecules to treat pre-eclampsia that we are aware of.

The Translational Obstetrics Group at Melbourne University has generated strong preclinical evidence suggesting esomeprazole as one of the proton pump inhibitors may have potent actions giving it significant potential as a treatment for pre-eclampsia

Proton pump inhibitors have been commonly used in pregnancy to treat gastroesophageal reflux disorders and more serious gastrointestinal complications like Helicobacter pylori-infection, peptic and duodenal ulcers and Zollinger-Ellison syndrome.

Esomeprazole counters three key steps in pre-eclampsia pathogenesis, by up-regulating heme oxygenase-1 ( strongly decreasing the release of antiangiogenic factors Soluble Fms Like Tyrosine Kinase -1 and soluble endoglin and quenching endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 28 + 0 weeks and 31 + 6 weeks
* Estimated fetal weight by ultrasound between 500 gm and 1800 gm (if gestation is not certain).
* Singleton pregnancy.
* The patient will be managed with expectant management.

Exclusion Criteria:

* Patient is unable or unwilling to give consent
* Established fetal compromise that necessitates delivery.
* The presence of any of the following at presentation:

  * Eclampsia.
  * Severe hypertension.
  * Cerebrovascular event as an ischaemic or haemorrhagic stroke.
  * Renal impairment.
  * Signs of left ventricular failure which include pulmonary oedema.
  * Disseminated intravascular coagulation (DIC)
  * Haemolysis, elevated liver enzymes and low platelets (HELLP syndrome)
  * Fetal distress on cardiotocography
* Contra-indications for expectant management of pre-eclampsia
* Current use of a proton pump inhibitor
* Contraindications to the use of a proton pump inhibitor
* Previous hypersensitivity reaction to a proton pump inhibitor

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 205 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Number of women who develop HELLP syndrome | 1 month
The change in serum level of sFlt-1 and endoglin before the start of treatment and at termination of pregnancy | 2 weeks

SECONDARY OUTCOMES:
Prolongation of gestation measured from the time of enrollment to the time of delivery | 2 weeks
The side effects of the drugs | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abbas, MD, Study Director — Assiut University
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cluver CA, Walker SP, Mol BW, Theron GB, Hall DR, Hiscock R, Hannan N, Tong S. Double blind, randomised, placebo-controlled trial to evaluate the efficacy of esomeprazole to treat early onset pre-eclampsia (PIE Trial): a study protocol. BMJ Open. 2015 Oct 28;5(10):e008211. doi: 10.1136/bmjopen-2015-008211. PMID 26510725
- [Background] Lagana AS, Favilli A, Triolo O, Granese R, Gerli S. Early serum markers of pre-eclampsia: are we stepping forward? J Matern Fetal Neonatal Med. 2016 Sep;29(18):3019-23. doi: 10.3109/14767058.2015.1113522. Epub 2015 Nov 23. PMID 26512423
- [Background] Baumann MU, Bersinger NA, Mohaupt MG, Raio L, Gerber S, Surbek DV. First-trimester serum levels of soluble endoglin and soluble fms-like tyrosine kinase-1 as first-trimester markers for late-onset preeclampsia. Am J Obstet Gynecol. 2008 Sep;199(3):266.e1-6. doi: 10.1016/j.ajog.2008.06.069. PMID 18771978